## **Title**

Surgical Therapy and Survival in Young Patients with Stage I-II Hepatocellular Carcinoma: A Retrospective Cohort Study

## Study Protocol and Statistical Analysis Plan

NCT04820712

From September 1, 2020 to September 30, 2017, complete the preparation for the study and obtain access to the public database From October 1, 2020 to October 31, 2020, download data from public database and analyze data

From November 1, 2020 to November 30, 2020, writing paper
From December 1, 2020 to December 31, 2020, thesis revision
From January 1, 2021 to now, make a comprehensive summary,
complete the final report, identify the achievements, and publish one
paper

## **Description of informed consent form**

The SEER data contain no identifiers and are publicly available for studies of cancer-based epidemiology and survival analysis. Therefore, the current study was deemed to be exempt from Institutional Review Board approval and the need for informed consent was waived.